CLINICAL TRIAL: NCT04382456
Title: An Exploratory Pilot Study to Evaluate the Impact of Alpinia Acacia Gum on Microbiome and Bowel Function in Subjects With Chronic Constipation
Brief Title: Evaluation of Acacia Gum on Microbiome and Bowel Function in Participants With Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alpinia Laudanum GmbH (Other)
Collaborators: BioTeSys GmbH (Other)
Responsible Party: Sponsor
Organization: Alpinia Laudanum Institute of Phytopharmaceutical Sciences AG (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BTS1416/19
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-08

CONDITIONS: Constipation
Keywords: Acacia gum; gummi arabicum; microbiome; short chain fatty acids; SCFA; stool frequency; stool consitency
MeSH Terms: conditions — Constipation | interventions — Gum Arabic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acacia gum (Experimental)
  Interventions: Dietary Supplement: acacia gum

INTERVENTIONS:
Dietary Supplement: acacia gum — Two sachets (à 5 g) in the morning and two sachets in the evening, reconstituted in 120 ml water and stirred until fully dissolved to be taken 10 minutes before meals.

SUMMARY:
Proof of concept study to investigate the impact of a food supplement consisting of Acacia gum on changes of gut microbiota and production of short chain fatty acids. Additionally, safety, tolerability and parameters of bowel function (stool frequency, stool consistency and gastrointestinal symptoms) will be assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without clinical diagnosed diseases with relevant effect on the gastrointestinal system or on visceral motility
* Constipation defined as an average of 2 - 3 stools per week (which needs to be confirmed during a prospective run-in phase)
* At least one of the following criteria:

  * straining during more than 25% of defecations
  * lumpy or hard stools (Bristol Stool Form Scale 1 or 2) present more than 25% of defecations
  * sensation of incomplete evacuation in more than 25% of defecations
  * sensation of anorectal obstruction/ blockage in more than 25% of defecations
  * manual manoeuvre to facilitate more than 25% of defecations (such as digital evacuation or support from pelvic floor)
* Criteria of constipation for at least the previous 3 months
* BMI 18.5 - 30 kg/m2
* Stable body weight (+/- 5%) in the last 3 months (self-reported)
* Willing to maintain normal background dietary habits & physical activity levels throughout the study period
* Written consent to participate in the study

Exclusion Criteria:

* Relevant history or presence of any severe medical disorder, potentially interfering with this study in the investigator's judgement (e.g. mal absorption, food intolerance or allergy, chronic gastro-intestinal diseases (e.g. Morbus Crohn, Colitis Ulcerosa), chronic kidney or liver disease, severe depression, immunological disorders, severe cardiovascular disease, diabetes, acute malignant disease within last 3 years except basal cell carcinoma of the skin)
* Prior abdominal surgery which may present a risk for the subject or confound the study results (according to the investigator's opinion)
* Currently (or in the last 3 months) suffering from significant stress, anxiety or depression which, in the subjects opinion, interferes with normal daily life (e.g. has the subject missed days of work due to these conditions) and/or which could be responsible for gastrointestinal problems
* Exclusively vegan or vegetarian diet (high fiber content)
* Regular laxative use at least once per week
* Use of hypolipidaemic drugs (e.g. statins, fibrates, resins, ezetimibe, niacin)
* Subject under prescription for medication or taking dietary supplements possibly interfering with this study (such as anti-spasmodic, laxatives and anti-diarrheic drugs or other digestive auxiliaries, use of PPIs, bismuth salts and/or H2-antagonists, fibers etc.) within 2 weeks prior to study start or during the study; Stable medication (more than 3 months) for hypertension or thyroid gland is allowed.
* Use of pre- and probiotic supplements
* Subjects consuming

  * food or drinks claimed as 'probiotic', or 'prebiotic more than once weekly
  * food or drinks claimed as 'rich in fiber' (including specific milk products) more than 3 times per week
  * more than 3 portions of fruits and vegetables (sum) per day
* Smoker
* Intake of antibiotics in the last 4 weeks
* Pregnancy or breastfeeding (also exclude recent pregnancy in the last 3 months). A pregnancy test will be conducted during screening and visits 1 - 3.
* Currently or recently (within 3 months of study entry) taking any medication, which in the opinion of the investigator, could interfere with the outcome of the study, e.g. opioids, anti-psychotics

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Gut microbiota | day 1, day 43 and day 71
  Composition and diversity (Shannon index), Lactobacillogenic and bifidogenic level, Distribution of bacterial taxa at the phylum, family and genus level, Shifts of specific bacterial taxa

SECONDARY OUTCOMES:
Stool frequency | day -14 (run-in phase) until day 70 (end of follow up)
  frequency per week will be assessed via diary
Stool consitency | day -14 (run-in phase) until day 70 (end of follow up)
  consistency will be assessed via Bristol Stool Form Scale
Gastrointestinal symptoms | day -14 (run-in phase) until day 70 (end of follow up)
  Global Gastrointestinal Discomfort Assessment (PAC-SYM), single gastrointestinal symptoms (flatulence, rumbling (i.e. borborygmi)), layative use
Blood biomarker | day 1, day 43 and day 71
  Lipid profile (total, HDL- and LDL- cholesterol and triglycerides) Blood glucose Electrolytes and minerals (plasma sodium, potassium and calcium) SCFA (short chain fatty acids) (optional) Cytokines: IL-10 & IL-6 (optional)
Stool biomarker | day 1, day 43 and day 71
  SCFA (short chain fatty acids) Zonulin Calprotectin (optional) Secretory IgA (optional) Beta-defensin (optional) Bile acids (optional) Nitric oxide (optional)

CONTACTS AND LOCATIONS:
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany